CLINICAL TRIAL: NCT01087502
Title: A Phase III, Randomised, Double-blind, Placebo-controlled Parallel Group Safety and Efficacy Study of Linagliptin (5 mg Administered Orally Once Daily) Over 12 Weeks Followed by a 40 Week Double-blind Extension Period (Placebo Patients Switched to Glimepiride) in Drug Naive or Previously Treated Type 2 Diabetic Patients With Moderate to Severe Renal Impairment and Insufficient Glycaemic Control
Brief Title: Safety and Efficacy of Linagliptin in Type-2-diabetes Mellitus Patients With Moderate to Severe Renal Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.64; 2009-016971-31 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; Linagliptin

ARMS (3):
- Linagliptin (Experimental): 52 weeks treatment
  Interventions: Drug: Placebo; Drug: Linagliptin
- Placebo (Placebo Comparator): First 12 weeks of treatment
  Interventions: Drug: Placebo
- Glimepiride (Active Comparator): Placebo patients switch to glimepiride after 12 weeks (40 weeks treatment)
  Interventions: Drug: Glimepiride; Drug: Placebo

INTERVENTIONS:
Drug: Glimepiride — 1-4 mg daily after 12 weeks
  Arms: Glimepiride
Drug: Placebo — Placebo mach to 5 mg linagliptin first 12 weeks of treatment once daily
  Arms: Placebo
Drug: Placebo — Placebo maching Glimepiride 1-4 mg after 12 weeks of treatment
  Arms: Linagliptin
Drug: Placebo — Placebo mach to 5 mg linagliptin once daily after 12 weeks
  Arms: Glimepiride
Drug: Linagliptin — 5 mg once daily
  Arms: Linagliptin

SUMMARY:
The objective of the current study is to investigate the efficacy, safety and tolerability of linagliptin (5 mg / once daily) compared to placebo given over 12 weeks in drug naive or previously treated type 2 diabetic patients with moderate to severe renal impairment and insufficient glycaemic control. In addition safety in this patient population with longer term (40 week) treatment in comparison to sulfonylurea drug (glimepiride).

ELIGIBILITY:
Inclusion criteria:

1. Type 2 diabetes mellitus
2. GFR<60 ml/min
3. HbA1c >=7.0% to <= 10%
4. Age >= 18 years
5. BMI <=45 kg/m2
6. Signed and dated written informed consent

Exclusion criteria:

1. Myocardial infarction, stroke or TIA within 3 months prior to informed consent
2. Renal impairment requiring dialysis
3. Bariatric surgery
4. Impaired hepatic function
5. Treatment with glitazones, GLP-1 analogues, DPP-4 inhibitors
6. Treatment with anti-obesity drugs
7. Treatment with SU, glinides and metformin 8 weeks prior to informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2010-03; Primary Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (52):
- United States (16):
  - 1218.64.10007 Boehringer Ingelheim Investigational Site, Chula Vista, California
  - 1218.64.10018 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 1218.64.10016 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 1218.64.10015 Boehringer Ingelheim Investigational Site, Boise, Idaho
  - 1218.64.10002 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1218.64.10004 Boehringer Ingelheim Investigational Site, Flint, Michigan
  - 1218.64.10006 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 1218.64.10003 Boehringer Ingelheim Investigational Site, The Bronx, New York
  - 1218.64.10013 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1218.64.10020 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1218.64.10008 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1218.64.10009 Boehringer Ingelheim Investigational Site, Arlington, Texas
  - 1218.64.10005 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1218.64.10011 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1218.64.10014 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1218.64.10010 Boehringer Ingelheim Investigational Site, Tacoma, Washington
- Australia (5):
  - 1218.64.61005 Boehringer Ingelheim Investigational Site, Gosford, New South Wales
  - 1218.64.61001 Boehringer Ingelheim Investigational Site, Liverpool, New South Wales
  - 1218.64.61002 Boehringer Ingelheim Investigational Site, St Leonards, New South Wales
  - 1218.64.61003 Boehringer Ingelheim Investigational Site, Adelaide, South Australia
  - 1218.64.61004 Boehringer Ingelheim Investigational Site, Reservoir, Victoria
- Canada (7):
  - 1218.64.20008 Boehringer Ingelheim Investigational Site, Corunna, Ontario
  - 1218.64.20005 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1218.64.20007 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1218.64.20002 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1218.64.20009 Boehringer Ingelheim Investigational Site, Stayner, Ontario
  - 1218.64.20004 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1218.64.20003 Boehringer Ingelheim Investigational Site, Point Claire, Quebec
- Finland (3):
  - 1218.64.35804 Boehringer Ingelheim Investigational Site, Kokkola
  - 1218.64.35803 Boehringer Ingelheim Investigational Site, Oulu
  - 1218.64.35801 Boehringer Ingelheim Investigational Site, Turku
- Israel (6):
  - 1218.64.97204 Boehringer Ingelheim Investigational Site, Ashkelon
  - 1218.64.97207 Boehringer Ingelheim Investigational Site, Giv‘atayim
  - 1218.64.97203 Boehringer Ingelheim Investigational Site, Haifa
  - 1218.64.97201 Boehringer Ingelheim Investigational Site, Jerusalem
  - 1218.64.97202 Boehringer Ingelheim Investigational Site, Nahariya
  - 1218.64.97206 Boehringer Ingelheim Investigational Site, Tel Aviv
- Japan (8):
  - 1218.64.81005 Boehringer Ingelheim Investigational Site, Asahi, Chiba
  - 1218.64.81006 Boehringer Ingelheim Investigational Site, Isesaki, Gunma
  - 1218.64.81001 Boehringer Ingelheim Investigational Site, Meguro-ku, Tokyo
  - 1218.64.81008 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1218.64.81007 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1218.64.81002 Boehringer Ingelheim Investigational Site, Shinjyuku-ku,Tokyo
  - 1218.64.81004 Boehringer Ingelheim Investigational Site, Suita, Osaka
  - 1218.64.81003 Boehringer Ingelheim Investigational Site, Suwa, Nagano
- 1218.64.64001 Boehringer Ingelheim Investigational Site, Otahuhu Auckland, New Zealand
- Slovakia (4):
  - 1218.64.42102 Boehringer Ingelheim Investigational Site, Bratislava
  - 1218.64.42107 Boehringer Ingelheim Investigational Site, Košice
  - 1218.64.42109 Boehringer Ingelheim Investigational Site, Nitra
  - 1218.64.42108 Boehringer Ingelheim Investigational Site, Trenčín
- Sweden (2):
  - 1218.64.46002 Boehringer Ingelheim Investigational Site, Härnösand
  - 1218.64.46003 Boehringer Ingelheim Investigational Site, Helsingborg

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 241 patients were randomised to treatment with linagliptin 5mg (n=118) or placebo/glimepiride (n=123). All randomised patients were treated. For the final analysis, one study site was excluded due to serious non-compliance resulting in 122 patients in the placebo/glimepiride group and 113 patients in the linagliptin group.
Groups:
- Placebo/Glimepiride: Patients randomized to receive treatment with matching placebo for 12 weeks and then switch to glimepiride for further 40 weeks.
- Linagliptin 5 mg: Patients randomized to receive treatment with Linagliptin 5mg
Period: Up to Interim Analysis (Week 12)
Arm/Group | Placebo/Glimepiride | Linagliptin 5 mg
Started | 123 | 118
Completed | 114 | 110
Not Completed | 9 | 8
Not completed — Adverse Event | 5 | 4
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Other reason not described above | 1 | 2
Period: Up to Final Analysis (Week 52)
Arm/Group | Placebo/Glimepiride | Linagliptin 5 mg
Started | 123 | 118
Completed | 90 | 95
Not Completed | 33 | 23
Not completed — Adverse Event | 17 | 10
Not completed — Lack of Efficacy | 1 | 2
Not completed — Protocol Violation | 4 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Study site excluded from analysis | 1 | 5
Not completed — Other reason not described above | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Glimepiride | Linagliptin 5 mg | Total
Number analyzed (Participants) | 122 | 113 | 235
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age Continuous for patient set up to 52 weeks
  Years | 65.9 (9.4) | 67.3 (9.2) | 66.6 (9.3)
Age, Continuous [Mean (Standard Deviation); unit: years] — Age Continuous for patient set up to 12 weeks (N=123, 118, 241)
  years | 65.6 (10.0) | 66.9 (9.4) | 66.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender for patient set up to 52 weeks.
  Participants
    Female | 43 | 43 | 86
    Male | 79 | 70 | 149
Gender [Number; unit: participants] — Gender for patient set up to 12 weeks (N=123, 118, 241)
  participants
    Female | 43 | 44 | 87
    Male | 80 | 74 | 154
Body mass index (BMI) continuous [Mean (Standard Deviation); unit: kg/m^2] — BMI for patient set up to 52 weeks.
  kg/m^2 | 31.97 (6.28) | 32.22 (5.99) | 32.09 (6.13)
Body mass index (BMI) continuous [Mean (Standard Deviation); unit: kg/m^2] — BMI for patient set up to 12 weeks (N=123, 118, 241)
  kg/m^2 | 31.93 (6.27) | 32.20 (6.13) | 32.06 (6.19)
Glycosylated Hemoglobin A1 (HbA1c) [Mean (Standard Deviation); unit: Percent] — HbA1c based on Full analysis set (FAS) up to 52 weeks (N=120, 113, 233)
  Percent | 8.03 (0.94) | 8.08 (0.89) | 8.05 (0.91)
Glycosylated Hemoglobin A1 (HbA1c) [Mean (Standard Deviation); unit: Percent] — HbA1c based on Full analysis set (FAS) up to 12 weeks (N=121, 117, 238)
  Percent | 8.02 (0.94) | 8.08 (0.88) | 8.05 (0.91)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — FPG based on Full analysis set (FAS) up to 52 weeks (N=120, 113, 233)
  mg/dL | 149.7 (53.1) | 155.3 (45.6) | 152.4 (49.6)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — FPG based on FAS up to 12 weeks (N=121, 117, 238)
  mg/dL | 149.3 (53.0) | 154.4 (46.1) | 151.8 (49.7)
eGFR based on Modification of Diet in Renal Disease (MDRD) formula [Number; unit: Participants] — eGFR based on FAS up to 52 weeks (N=122, 113, 235). eGFR means Estimated glomerular filtration rate.
  Participants
    >=90 (normal renal function) | 0 | 0 | 0
    60 to <90 (mild renal impairment) | 4 | 6 | 10
    30 to <60 (moderate renal impairment) | 73 | 72 | 145
    <30 (severe or endstage renal impairment) | 45 | 35 | 80
eGFR based on Modification of Diet in Renal Disease (MDRD) formula [Number; unit: participants] — eGFR based on FAS up to 12 weeks (N=123, 118, 241). eGFR means Estimated glomerular filtration rate.
  participants
    >=90 (normal renal function) | 0 | 0 | 0
    60 to <90 (mild renal impairment) | 5 | 6 | 11
    30 to <60 (moderate renal impairment) | 73 | 76 | 149
    <30 (severe or endstage renal impairment) | 45 | 36 | 81

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline to Week 12
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 12 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c, renal function impairment and prior use of antidiabetic agents.
Time Frame: Baseline and week 12
Population: FAS consisting of all randomised patients who were treated with at least one dose of study drug, had a baseline, and at least 1 on-treatment HbA1c measurement. Last observation carried forward (LOCF) was used as the imputation rule.
  Results for primary endpoint below are the ones reproduced without patients from the excluded study site.
Measure: Mean (Standard Error); unit: Percent
Groups:
- Placebo: Patients randomized to receive treatment with matching placebo for 12 weeks and then switch to glimepiride for further 40 weeks.
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 120 | 113
Percent | -0.11 (0.11) | -0.53 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.42, 95% CI [-0.60 to -0.24], Standard Error of Mean 0.09

2. Secondary Outcome: HbA1c Change From Baseline Over Time
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the HbA1c percent over time minus the baseline HbA1c percent. This outcome measure only provides descriptive statistics without any modelling.
Time Frame: Baseline, week 4, week 8, week 12, week 16, week 20, week 24, week 28, week 34, week 40, week 46, week 52
Population: FAS. Last observation carried forward (LOCF) was used as the imputation rule. Results do not contain data of patients from the excluded study site.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Placebo/Glimepiride | Linagliptin 5 mg
Number analyzed (Participants) | 120 | 113
Percent
  Week 4 (N=120, 113) | -0.08 (0.42) | -0.29 (0.35)
  Week 8 (N=120, 113) | -0.09 (0.68) | -0.47 (0.49)
  Week 12 (N=120, 113) | -0.08 (0.79) | -0.50 (0.59)
  Week 16 (N=120, 113) | -0.31 (0.84) | -0.47 (0.61)
  Week 20 (N=120, 113) | -0.48 (0.88) | -0.48 (0.63)
  Week 24 (N=120, 113) | -0.51 (0.93) | -0.52 (0.66)
  Week 28 (N=120, 113) | -0.47 (0.93) | -0.50 (0.68)
  Week 34 (N=120, 113) | -0.37 (0.93) | -0.45 (0.69)
  Week 40 (N=120, 113) | -0.23 (0.95) | -0.42 (0.73)
  Week 46 (N=120, 113) | -0.24 (0.96) | -0.40 (0.75)
  Week 52 (N=120, 113) | -0.25 (0.92) | -0.40 (0.77)

3. Secondary Outcome: Fasting Plasma Glucose (FPG) Change From Baseline to Week 12
Description: This change from baseline reflects the Week 12 FPG minus the baseline FPG. Means are treatment-adjusted for baseline HbA1c, baseline FPG and prior use of insulin, week repeated within patient and week by treatment interaction.
Time Frame: Baseline and week 12
Population: One patient in the Placebo/Glimepiride arm and one patient in the Linagliptin arm without FPG on-treatment value. Results do not contain data of patients from the excluded study site.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo/Glimepiride | Linagliptin 5 mg
Number analyzed (Participants) | 119 | 112
mg/dL | 9.53 (8.01) | 0.24 (7.71)
Statistical Analysis 1: Comparison: Placebo/Glimepiride vs Linagliptin 5 mg; Test type: Superiority or Other; p = 0.1602, ANCOVA; Mean Difference (Final Values) = -9.29, 95% CI [-22.28 to 3.7], Standard Error of Mean 6.59

4. Secondary Outcome: Fasting Plasma Glucose (FPG) Change From Baseline Over Time
Description: This change from baseline reflects the FPG over time minus the baseline FPG. This outcome measure only provides descriptive statistics without any modelling.
Time Frame: Baseline, week 4, week 8, week 12, week 20, week 24, week 28, week 34, week 40, week 46, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo/Glimepiride | Linagliptin 5 mg
Number analyzed (Participants) | 119 | 112
mg/dL
  Week 4 (N=119, 112) | 9.80 (54.94) | -10.55 (45.80)
  Week 8 (N=119, 112) | 8.96 (53.30) | -11.25 (52.32)
  Week 12 (N=119, 112) | 6.23 (58.20) | -6.26 (52.59)
  Week 20 (N=119, 112) | -9.66 (60.60) | -5.92 (57.68)
  Week 24 (N=119, 112) | -8.83 (54.84) | -12.78 (62.29)
  Week 28 (N=119, 112) | -9.67 (58.31) | -9.31 (61.01)
  Week 34 (N=119, 112) | -9.95 (58.47) | -2.78 (64.55)
  Week 40 (N=119, 112) | -0.75 (61.94) | -2.69 (68.43)
  Week 46 (N=119, 112) | -2.64 (60.83) | -2.03 (71.30)
  Week 52 (N=119, 112) | -3.10 (58.27) | 3.09 (69.03)

5. Secondary Outcome: Percentage of Patients With HbA1c <7.0%
Description: The percentage of patients with an HbA1c value below 7% at week 12 and week 52 were calculated for each treatment arm. If a patient did not have an HbA1c value at week 12 or 52 respectively, they were considered a failure, so HbA1c above 7%.
Time Frame: Baseline, week 12 and week 52
Population: FAS with baseline HbA1c >=7% and non-completers considered as failure imputation (NCF). Results after Week 12 include patients from the excluded study site.
Measure: Number; unit: percentage of patients
Arm/Group | Placebo/Glimepiride | Linagliptin 5 mg
Number analyzed (Participants) | 110 | 108
percentage of patients
  Week 52 (N=110, 104) | 11.8 | 22.1
  Week 12 (N=110, 108) | 9.1 | 19.4

6. Secondary Outcome: Percentage of Patients With HbA1c <6.5%
Description: The percentage of patients with an HbA1c value below 6.5% at week 12 and week 52 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 12 or 52 respectively they were considered a failure, so HbA1c above 6.5%.
Time Frame: Baseline, week 12 and week 52
Population: FAS with baseline HbA1c >=6.5% and non-completers considered as failure imputation (NCF). Results after Week 12 include patients from the excluded study site.
Measure: Number; unit: percentage of patients
Arm/Group | Placebo/Glimepiride | Linagliptin 5 mg
Number analyzed (Participants) | 120 | 115
percentage of patients
  Week 52 (N=119, 111) | 6.7 | 9.9
  Week 12 (N=120, 115) | 5.0 | 6.1

7. Secondary Outcome: Percentage of Patients Who Have a HbA1c Lowering by at Least 0.5%
Description: The percentage of patients with an HbA1c reduction of ≥0.5% at week 12 and week 52 from baseline was calculated for each treatment arm. If a patient did not have an HbA1c value at week 12 or 52 respectively they were considered a failure, so HbA1c reduction less than 0.5%.
Time Frame: Baseline, week 12 and week 52
Population: FAS with non-completers considered as failure imputation (NCF). Results after Week 12 include patients from the excluded study site.
Measure: Number; unit: percentage of patients
Arm/Group | Placebo/Glimepiride | Linagliptin 5 mg
Number analyzed (Participants) | 121 | 117
percentage of patients
  Week 52 (N=120, 113) | 23.3 | 34.5
  Week 12 (N= 121, 117) | 24.0 | 49.6

8. Secondary Outcome: Plasma Concentration of Linagliptin at Trough
Description: Trough levels of concentration of Linagliptin in plasma.
Time Frame: Week 12, 24 and 52
Population: FAS original results (OR). Original results analysis means that data is analyzed exactly as observed, values after rescue medication are not set to missing and no imputation rule is applied for replacing the missing values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nmol/L
Arm/Group | Linagliptin 5 mg
Number analyzed (Participants) | 113
Nmol/L
  Week 12 (N=103) | 7.77 (36.43)
  Week 24 (N=103) | 7.62 (41.04)
  Week 52 (N=105) | 5.94 (107.40)

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Placebo/Glimepiride | Linagliptin 5 mg
Serious Adverse Events (participants affected / at risk) | 36/122 | 28/113
Other Adverse Events (participants affected / at risk) | 110/122 | 95/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Glimepiride (N=122) | Linagliptin 5 mg (N=113)
Pneumonia (Infections and infestations) | 2 | 3
Cellulitis (Infections and infestations) | 3 | 0
Gastroenteritis (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 2 | 0
Acarodermatitis (Infections and infestations) | 0 | 1
Gas gangrene (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Endocarditis enterococcal (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Fluid retention (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Brachial plexopathy (Nervous system disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 5 | 4
Acute myocardial infarction (Cardiac disorders) | 3 | 0
Angina pectoris (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 2
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Chest pain (General disorders) | 4 | 1
Oedema peripheral (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Glimepiride (N=122) | Linagliptin 5 mg (N=113)
Nasopharyngitis (Infections and infestations) | 18 | 21
Upper respiratory tract infection (Infections and infestations) | 10 | 11
Urinary tract infection (Infections and infestations) | 8 | 8
Bronchitis (Infections and infestations) | 8 | 7
Influenza (Infections and infestations) | 7 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 85 | 67
Hyperglycaemia (Metabolism and nutrition disorders) | 20 | 20
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 8
Headache (Nervous system disorders) | 8 | 4
Dizziness (Nervous system disorders) | 7 | 6
Hypertension (Vascular disorders) | 6 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Constipation (Gastrointestinal disorders) | 12 | 6
Diarrhoea (Gastrointestinal disorders) | 7 | 6
Vomiting (Gastrointestinal disorders) | 3 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 8
Oedema peripheral (General disorders) | 9 | 3
Fall (Injury, poisoning and procedural complications) | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.